CLINICAL TRIAL: NCT01161784
Title: The Effects of a Probiotic Fermented Milk on Functional Constipation in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Collaborators: University of Malaya (Other); National University of Malaysia (Other)
Responsible Party: Prof. Dr. Fatimah Arshad, International Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMU RO52/2009
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Constipation
Keywords: Functional constipation; Probiotic; Probiotic microorganism; Lactobacillus casei Shirota (LcS)
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrient drink (Placebo Comparator)
  Interventions: Dietary Supplement: Nutrient drink
- Probiotics (Experimental)
  Interventions: Dietary Supplement: Probiotics fermented milk

INTERVENTIONS:
Dietary Supplement: Probiotics fermented milk — 80ml fermented milk containing min. 30 billion live L. casei Shirota strain, administered orally once a day for 4 weeks
  Arms: Probiotics
Dietary Supplement: Nutrient drink — 80ml fermented milk without L. casei Shirota strain, administered orally once a day for 4 weeks
  Arms: Nutrient drink

SUMMARY:
The purpose of this study is to determine the effects of daily consumption for 4 weeks of a fermented milk drink containing a live probiotic microorganism, Lactobacillus casei strain Shirota (LcS) compared to a placebo without LcS, among adults with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with functional constipation based on ROME II criteria
* Has a constipation severity score (Chinese Constipation Questionnaire or CCQ score) of at least 5, which is the cut-off point for constipated subjects (Chan et al, 2005)
* Free of any cardiovascular related diseases, diabetes, cancer, neurological diseases or any other serious illness, not physically or mentally handicapped
* Living in Klang Valley, with no pre-determined plans to be out of town for one week or longer during scheduled intervention period

Exclusion Criteria:

* Body Mass Index of less than 16, or 30 and above
* Pregnant
* Regular ingestion of probiotic products within the preceding four weeks
* Regular use of laxatives (average once a week or more)
* Intake of anticholinergics medications or medications against diarrhea or antibiotics in the preceding 1 month
* Persons with milk protein allergy
* Persons with constipation of organic or neurological origin based on health screening
* Persons with alarm features as assessed by physician during health screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Constipation severity score which measures overall signs and symptoms of constipation using the 'Chinese Constipation Questionnaire' or CCQ (Chan et al, 2005) | 4 weeks
  Constipation severity score is patient self-assessment of 6 signs and symptoms of constipation:
  1. Severity of false alarms
  2. Frequency of less than 3 defecations / week
  3. Severity of sensation of incomplete bowel movement
  4. Severity of lumpy or hard stools
  5. Severity of bloating
  6. Frequency of laxative use
Frequency of bowel movement | 4 weeks

SECONDARY OUTCOMES:
Stool consistency based on modified Bristol Stool scale | 4 weeks
  Stool consistency is self-assessed by subjects as Type 1,2,3,4 or 5.
Stool output quantity estimations | 4 weeks
  Stool output is estimated by subjects visually based on comparison to size of a standard ping pong ball.

CONTACTS AND LOCATIONS:
Locations (1):
- International Medical University, Kuala Lumpur, Kuala Lumpur, Malaysia